CLINICAL TRIAL: NCT02225093
Title: A Phase 1 Open-label Study to Evaluate the Effect of Multiple Doses of Enzalutamide on the Pharmacokinetics of Substrates for CYP1A2 and CYP2D6 in Male Subjects With Prostate Cancer
Brief Title: A Study to Evaluate How Daily Dosing With Enzalutamide Affects the Metabolism of Caffeine and Dextromethorphan in Men With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 9785-CL-0406
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Pharmacokinetics of Dextromethorphan; Pharmacokinetics of Caffeine; Prostate Cancer
Keywords: Safety; Dextromethorphan; CYP2D6; Phase 1; Prostate cancer; CYP1A2; Pharmacokinetics; Drug-drug interactions; Caffeine; Enzalutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Caffeine; Dextromethorphan; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1:Caffeine, Dextromethorphan and Enzalutamide (Experimental): 1-sequence crossover here
  Interventions: Drug: Caffeine; Drug: Dextromethorphan; Drug: Enzalutamide; Drug: Enzalutamide Placebo to Match (PTM)

INTERVENTIONS:
Drug: Caffeine — Oral
  Other Names: CYP1A2 substrate
Drug: Dextromethorphan — Oral /.L
  Other Names: CYP2D6 substrate
Drug: Enzalutamide — Oral
  Other Names: Xtandi; MDV3100; ASP9785
Drug: Enzalutamide Placebo to Match (PTM) — Oral

SUMMARY:
This study evaluates how once daily enzalutamide affects the metabolism of caffeine and dextromethorphan in men with prostate cancer by measuring concentrations of these drugs and their metabolites in plasma.

DETAILED DESCRIPTION:
This is an open-label, fixed-sequence, crossover drug-drug interaction study in subjects with prostate cancer.

Screening takes place between Day -28 and Day -7, and subjects are admitted to the clinic on Day -1 where they remain until Day 4.

On Day 1, they receive a single oral cocktail containing caffeine and dextromethorphan plus a dose of enzalutamide placebo in order to assess possible effects of excipients of the enzalutamide formulation. On Days 1 to 3 blood samples for pharmacokinetic (PK) assessment are collected. From Days 4 to 54, (or Day 55 if the subject rolls over into the extension study) the subjects take a daily oral dose of enzalutamide. On Day 28, the subjects return to the clinic where a plasma sample is taken to determine enzalutamide PK exposure. From Days 52 to 55 they are re-admitted to the clinic where a plasma sample is collected on Day 52 for enzalutamide PK exposure.On Day 53, subjects receive a single oral cocktail of caffeine and dextromethorphan concomitantly with enzalutamide. PK samples are collected from Days 53 to 55.

From Day 55 onwards, subjects experiencing clinical benefit may roll over into an extension study. Only subjects who enroll into the extension study continue to receive enzalutamide otherwise daily dosing with enzalutamide is discontinued on Day 54.

An End of Study Visit (ESV) takes place approximately 30 days (±7 days) after the last dose of enzalutamide.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male aged 18 years old or older (at screening) with histologically confirmed prostate cancer (all stages) for whom androgen deprivation therapy is indicated (except when indicated in a neoadjuvant/adjuvant setting). Subjects may be on ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue or have undergone prior bilateral orchiectomy at screening.
* Subject has progressive disease by prostate-specific antigen (PSA) or imaging.
* Subject has received no more than 2 prior chemotherapy regimens.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Male subject must use a condom if having sex with a pregnant woman.
* Male subject and their female spouse/partners who are of childbearing potential must use 2 acceptable methods of birth control starting at screening and continuing throughout the study period and for 3 months after final study drug administration.
* Subject has an estimated life expectancy of at least 6 months.

Exclusion Criteria:

* Subject has confirmed CYP2D6 poor metabolizer, or CYP2D6 ultrarapid metabolizer status based on genotyping analysis.
* Subject has known metastases in the liver or any hepatic disorder that could affect drug metabolism deemed clinically significant by the investigator after discussion with the sponsor.
* Subject has undergone major surgery within 4 weeks prior to day 1.
* Subject received treatment with chemotherapy within 4 weeks prior to enrollment (day 1 visit) or plans to initiate treatment with chemotherapy during the study.
* Subject uses concomitant medications that are potent inducers and/or inhibitors of CYP1A2, CYP2C8, CYP2D6, or CYP3A4.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10-02 (Actual); Primary Completion 2014-02-03 (Actual); Study Completion 2014-02-03 (Actual)

PRIMARY OUTCOMES:
PK measured by Pharmacokinetic parameter Maximum concentration (Cmax) | Day 1 and Day 53 (28 times)
  For the probe substrates (caffeine and dextromethorphan) in combination with enzalutamide PTM and in combination with enzalutamide.
PK measured by Pharmacokinetic parameter Area under the curve (AUC) from the time of dosing to the last measurable concentration (AUC0-t) | Day 1 and Day 53 (28 times)
  For the probe substrates (caffeine and dextromethorphan) in combination with enzalutamide PTM and in combination with enzalutamide.
PK measured by PK parameter area under the curve (AUC) from time 0 extrapolated to infinity (AUC0-inf) | Day 1 and Day 53 (28 times)
  For the probe substrates (caffeine and dextromethorphan) in combination with enzalutamide PTM and in combination with enzalutamide.

SECONDARY OUTCOMES:
PK measured by PK parameters tmax, terminal elimination half-life (t1/2), apparent total systemic clearance after oral dosing (CL/F), apparent volume of distribution during terminal elimination phase (Vz/F) and extrapolated AUC (%AUC) | Day 1 and Day 53 (28 times)
  Tmax is time to maximum concentration. These PK parameters will be measured for the probe substrates (caffeine and dextromethorphan) in combination with enzalutamide PTM and in combination with enzalutamide.
PK measured by PK parameters Cmax, AUC0-t, AUC0-inf, %AUC, tmax and t1/2 | Day 1 and Day 53 (28 times)
  For 1,7-dimethylxanthine (metabolite caffeine), dextrorphan (metabolite dextromethorphan).
PK measured by PK parameters Cmax, trough concentrations (Ctrough) at Days 28, 52, 53, 54 and 55, tmax, AUC during the time interval between consecutive dosing (AUCtau), CL/F (parent only) and peak-to-trough ratio (PTR) | Day 28 (± 1 day), and Days 52 to 55 (15 times)
  For Enzalutamide, N-desmethyl enzalutamide (M2) and sum of enzalutamide + M2.
Safety and tolerability measured by vital signs, adverse events, laboratory assessments and electrocardiogram | Screening (Day -28 to Day -7) to ESV (>153 times)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Arensia, Chisinau, Moldova

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=43